CLINICAL TRIAL: NCT06649266
Title: A Phase 2a, Multicentre Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of RBD1016 in Participants With Chronic Hepatitis D Virus Infection, Including a Randomised, Single Blinded, Placebo-controlled Exploratory Part
Brief Title: Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of RBD1016 in Participants With Chronic Hepatitis D
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ribocure Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC04T001
Record Dates: First submitted 2024-09-18; First posted 2024-10-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Hepatitis D
MeSH Terms: conditions — Hepatitis D, Chronic

STUDY DESIGN:
Intervention Model Description: Partly blinded, placebo-controlled clinical trial with an active and a deferred active group.
Masking Description: First part of the trial: All participants will be blinded to the trial treatment for the first 16 weeks after the first dose. Then, investigators and other clinic staff will be unblinded, i.e., they will know which treatment the participants receive at all times.
  Open-label extension part: additionally 3 doses of active IMP administered 12 weeks apart (site 01 only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Participants will receive RBD1016 (subcutaneous injections).
  Interventions: Drug: RBD1016
- Deferred active group (Other): Participants will receive 4 doses of placebo (subcutaneous injections) followed by RBD1016 (subcutaneous injections).
  Interventions: Drug: RBD1016; Drug: Placebo

INTERVENTIONS:
Drug: RBD1016 — RBD1016, active drug.
Drug: Placebo — Placebo that is identical in appearance and volume to the doses of active IMP.
  Arms: Deferred active group

SUMMARY:
The goal of this clinical trial is to learn if drug RBD1016 works to treat chronic hepatitis D virus infection in adults. It will also learn about the safety of drug RBD1016. The main questions it aims to answer are:

Does drug RBD106 reduce the HDV RNA levels? What medical problems may participants experience when taking drug RBD1016? Researchers will compare drug RBD1016 to a placebo to see if drug RBD1016 works to treat chronic hepatitis D.

Participants will:

Receive drug RBD1016 or a placebo several times throughout the trial. Visit the clinic once every 4-6 weeks for checkups and tests.

DETAILED DESCRIPTION:
This is a multicentre, randomised, partly blinded, placebo-controlled clinical trial to evaluate the efficacy, safety and pharmacokinetics (PK) of RBD1016 subcutaneous injections in participants with chronic HDV infection.

First part of the trial: There will be 2 treatment groups - an active group (n=10) and a deferred active group (n=5), with participants allocated randomly. In the active group, participants will receive RBD1016. In the deferred active group, participants will receive 4 doses of placebo followed by deferred treatment with doses of RBD1016.

Both groups will be on a stable nucleoside analogue (NA) treatment course during the trial . All participants will be blinded to the trial treatment for the 16 weeks after the first dose. Then, investigators and other clinic staff will be unblinded, i.e., they will know which treatment the participants receive at all times.

Open-label extension part (site 01 only): continued IMP-treatment with additionally 3 doses of IMP administered 12 weeks apart. This part of the trial is conducted to collect long-term safety data and further exploratory efficacy measures. Only participants who may benefit from continued treatment in the ,trial, according to the judgement of the investigator, will be eligible for the open-label extension part of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Male or female participant aged 18 to 65 years, inclusive.
3. Body mass index (BMI) ≥ 18 and ≤ 35 kg/m2 at the time of the screening visit.
4. Documented evidence of HDV infection in medical history, i.e., HDV antibodies (HDVAb) and/or HDV RNA positive test results within at least 6 months prior to screening.
5. Documented evidence of HBV infection in medical history, i.e., HBsAg and/or HBV DNA positive test results within at least 6 months prior to screening.
6. Documented absence of liver cirrhosis, defined as an LSM ≥ 10 kPa measured on FibroScan® elastography at screening.

Exclusion Criteria:

1. Laboratory results at screening as follows, or any clinically significant laboratory parameter outliers that may interfere with the evaluation of efficacy and/or safety in the trial, at the discretion of the Investigator:

   * α-fetoprotein (AFP) > 50 µg/L.
   * Albumin concentration < 3.0 g/dL.
   * International normalized ratio (INR) > 1.5.
   * Platelet count < 90 × 109/L.
   * Direct bilirubin > 2 × ULN, Gilbert syndrome excluded.
   * Creatinine concentration > 1.5 × ULN.
   * Creatinine clearance < 60 mL/min, according to the Cockcroft-Gault equation.
2. Positive result at screening for hepatitis C virus (HCV) and/or human immunodeficiency virus (HIV) and/or prior diagnosis of syphilis, acute hepatitis A and/or acute hepatitis E.
3. Prior diagnosis of other liver diseases of non-HBV or non-HDV aetiology, including autoimmune liver disease (e.g., autoimmune hepatitis, primary biliary cholangitis or primary sclerosing cholangitis), inherited metabolic liver disease (e.g., haemochromatosis, Wilson's disease, familial intrahepatic cholestasis), drug-induced liver disease and/or non alcoholic steatohepatitis (NASH) assessed as moderate or above, at the discretion of the Investigator.
4. Prior or current diagnosis of liver cirrhosis.
5. History of or active hepatic decompensation, e.g., ascites, variceal bleeding or hepatic encephalopathy, at the discretion of the Investigator.
6. History of organ transplantation, previous or concurrent HCC or imaging finding suggesting malignant liver lesions, at the discretion of the Investigator.
7. Signs of liver malignancy in abdominal ultrasound at screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Mean change (log10 value) vs. baseline in HDV RNA levels in plasma at end of trial (Week 60). | 60 weeks

SECONDARY OUTCOMES:
Frequency, intensity and seriousness of reported AEs, SAEs and AEs of special interest (AESIs) during the trial. | 60 weeks
  Number and percentage of participants with AEs, SAEs and AEs of interest. All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).
Mean change (log10 value) in HBsAg levels vs. baseline, at end of trial (Week 60). | 60 weeks
Proportion of participants with positive immunogenicity, measured as plasma concentrations of anti-drug antibodies (ADAs), at each evaluation time point up to end of the study at week 60. | 60 weeks
Mean maximum change (log10 value) in HDV RNA levels in plasma vs. baseline, at any timepoint during the study, and up to the end of study at Week 60. | Up to 60 weeks
  Mean maximum change refers to the average of the largest changes in HDV RNA levels.
Mean maximum change (log10 value) in HBsAg levels vs. baseline, at any timepoint during the study, and up to end of study at Week 60. | Up to 60 weeks
  Mean maximum change refers to the average of the largest changes in HBsAg levels.
For participants with HBsAg levels more than100 IU/mL at baseline: Proportion of participants with HBsAg levels ≤ 10 IU/mL at end of trial (Week 60). | 60 weeks
  Proportion of refers to the percentage or fraction of participants in the trial who meet the specified criteria.
Proportion of participants with undetectable HDV RNA (i.e., less than the limit of detection), or ≥ 2 log10 decrease in HDV RNA and alanine transaminase (ALT) normalisation, at end of trial (Week 60). | 60 weeks
  Proportion of refers to the percentage or fraction of participants in the trial who meet the specified criteria.
Proportion of participants with undetectable HDV RNA (i.e., less than the limit of detection) or ≥ 2 log10 decrease in HDV RNA at end of trial (Week 60). | 60 weeks
  Proportion of refers to the percentage or fraction of participants in the trial who meet the specified criteria.
Plasma concentrations of RBD1016. | 60 weeks

OTHER OUTCOMES:
Frequency, intensity and seriousness of reported AEs, SAEs and AEs of special interest | Week 60 to week 108
  Number and percentage of participants with reported AEs, SAEs and AEs of special interest. All reported AE terms will be coded using Medical Dictionary for Drug Regulatory Affairs (MedDRA).
Dynamic changes based on local lab measurements, of HDV RNA, HBsAg, HBsAb-status and HBV DNA levels | at each evaluation time point of the extension part of the trial up to end of trial extension (Week 108
  Dynamic changes based on local lab measurements, of HDV RNA, HBsAg, HBsAb-status and HBV DNA levels
Proportion of participants with undetectable HDV RNA (i.e, < limit of detection based on local lab measurement) | at any evaluation time point of the extension part of the trial.
  Proportion of participants with undetectable HDV RNA (i.e, < limit of detection based on local lab measurement)

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Medicinsk enhet för Infektionssjukdomar, Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Infektionskliniken, Danderyds sjukhus, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Undecided